CLINICAL TRIAL: NCT05363241
Title: Comparison of Genicular Nerve Denervation by Cooled Radiofrequency Using Classical and Revised Anatomical Targets for Pain Management of Osteoarthritis of the Knee Osteoarthritis: Clinical Study
Brief Title: Management of Knee Pain by Cooled Radiofrequency in Classical Anatomical Targets and Revised Targets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Alfenas (Other)
Collaborators: SINPAIN LTDA (Unknown)
Responsible Party: Principal Investigator, Rafaela Figueiredo Rodriques, Principal Investigator, Universidade Federal de Alfenas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5.354.533
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee; Pain, Chronic; Analgesia
Keywords: Knee Osteoarthritis; denervation of sensory nerves of the knee; classical targets; revised targets
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative group (CG) (No Intervention): The patients will receive standard pharmacological treatment (oral analgesics, intra-articular injection with corticosteroids) and physiotherapy for 6 months, where the end of the study occurs. After this period, the patient is guaranteed to undergo the cooled radiofrequency procedure, with medical indication.
- Radiofrequency cooled group with classical targets (CRF-CT) (Experimental): The patients will undergo the CRF procedure using the classical therapeutic targets (medial superior genicular nerve, lateral superior genicular nerve, medial inferior genicular nerve). So that patients do not know in which group of the study they are included, the probe will be placed in the aforementioned genicular nerves and also in the recurrent fibular nerve and in the infra-patellar branch of the saphenous nerve, but will not receive radiofrequency in the recurrent fibular nerve nor in the infra-patellar branch of the saphenous nerve, receiving radiofrequency only in the genicular nerves. Oral analgesics will be prescribed for the patient to use if necessary.
  Interventions: Procedure: Cooled radiofrequency in classical targets (CRF-CT)
- Radiofrequency cooled group with revised targets (CRF-RT) (Experimental): The patients will undergo the CRF procedure using the revised therapeutic targets (medial superior genicular nerve, lateral superior genicular nerve, medial inferior genicular nerve, recurrent fibular nerve and in the infra-patellar branch of the saphenous nerve). So that patients do not know in which group of the study they are included, the probe will be placed in all the aforementioned nerves and will receive radiofrequency in all of them. Oral analgesics will be prescribed for the patient to use if necessary.
  Interventions: Procedure: Cooled radiofrequency in revised targets (CRF-RT)

INTERVENTIONS:
Procedure: Cooled radiofrequency in classical targets (CRF-CT) — Participant will take Midazolam 2 mg as a sedative, and will be positioned on a fluoroscopy table in a supine posture, with a pillow under the knee allowing the knee in a slightly flexed position. The skin and subcutaneous tissues will be anesthetized with 2 mL of 1% lidocaine under sterile circumstances. Patients will undergo motor block tests, using 45 volts and 2 hertz, prior to the CRF itself, to ensure that no motor structures will be affected. If the motor test is negative, the CRF procedure will follow, using COOLIEF needles guided by fluoroscopy. A cooled technical chamber will be used, at a temperature of 60° and application for 150 seconds. The targets will be the genicular nerves superior medial, superior lateral, and inferior medial. The participant will not be able to follow the procedure.
  Arms: Radiofrequency cooled group with classical targets (CRF-CT)
Procedure: Cooled radiofrequency in revised targets (CRF-RT) — Participant will take Midazolam 2 mg as a sedative, and will be positioned on a fluoroscopy table in a supine posture, with a pillow under the knee allowing the knee in a slightly flexed position. The skin and subcutaneous tissues will be anesthetized with 2 mL of 1% lidocaine under sterile circumstances. Patients will undergo motor block tests, using 45 volts and 2 hertz, prior to the CRF itself, to ensure that no motor structures will be affected. If the motor test is negative, the CRF procedure will follow, using COOLIEF needles guided by fluoroscopy. A cooled technical chamber will be used, at a temperature of 60° and application for 150 seconds. The targets will be the genicular nerves superior medial, superior lateral, and inferior medial and recurrent fibular nerves and the infra-patellar branch of the saphenous nerve. The participant will not be able to follow the procedure.
  Arms: Radiofrequency cooled group with revised targets (CRF-RT)

SUMMARY:
Osteoarthritis (OA) is a chronic and progressive disease that results from characteristic pathological changes in the tissues of the entire joint, resulting in failure in the component parts. OA is one of the most common causes of disability in adults due to pain and altered joint function, impacting patients' quality of life. Treatment is based on decreasing pain and improving function, involving non-pharmacological, pharmacological, and surgical management. First-line treatment involves non-pharmacological and pharmacological measures. When OA is very advanced, total joint replacement surgery is recommended. However, for patients refractory to conservative treatment and unwilling or unable to undergo arthroplasty, few options remain. Recently, several studies involving minimally invasive procedures are being recommended. Among them is the cooled radiofrequency technique, causing neurotomy by thermal activity, thus reducing the patient's perception of pain. The classical therapeutic target for this technique are the genicular nerves of the knee. However, more recent studies have shown that these classical targets do not provide complete pain relief and have suggested new therapeutic targets, comprising besides the genicular nerves, the recurrent peroneal nerve and the infra-patellar branch of the saphenous nerve. In order to validate these revised targets, new studies need to be done. Therefore, the aim of the present study is to evaluate the efficacy of the cooled radiofrequency procedure using classical and revised targets, and to compare pain intensity, knee function, quality of life, analgesic consumption and adverse effects of both techniques.

Key words: Osteoarthritis of the knee. Sensory nerve denervation. Classical targets. Revised targets.

DETAILED DESCRIPTION:
The present clinical study will be prospective, randomized and double-blind (the principal investigator and the patients will be blinded; the interventional physicians will not be blinded).

Patients (n=60) from the Unified Health System of Brazil (SUS), seen at the Singular Alfenas Clinic, selected by the medical team, who meet all inclusion requirements, will be considered for this study; those who agree will sign the informed consent form.

After being selected, patients will undergo a test block on the genicular nerves and those who have an improvement of at least 50% will be eligible for the cooled radiofrequency procedure (CRF). Patients will be randomly divided into 3 groups (n=20 patients/group) by sort, made by an external researcher: a) conservative group (CG): patients will receive standard pharmacological treatment (oral analgesics, intra-articular injection with corticosteroids) and physiotherapy for 6 months, and after that period, the performance of the cooled radiofrequency procedure will be guaranteed, with medical indication; b) group cooled radiofrequency with classical targets (CRF-CT): patients will undergo the CRF procedure, using the classical therapeutic targets (medial superior genicular nerve, lateral superior genicular nerve, medial inferior genicular nerve and infra-patellar branch of the saphenous nerve).

In order that patients do not know in which group of the study they are included, the probe will be placed on the aforementioned genicular nerves as well as on the recurrent peroneal nerve and the the recurrent fibular nerve and the infra-patellar branch of the saphenous nerve, but will not receive radiofrequency in the recurrent fibular nerve nor in the infra-patellar branch of the saphenous nerve, receiving radiofrequency only in the genicular nerves; c) group cooled radiofrequency with revised targets (CRF-RT): patients will undergo the CRF procedure using the revised therapeutic targets (medial superior genicular nerve, lateral superior genicular nerve; medial inferior genicular nerve, fibular recurrent nerve and infra-patellar branch of the saphenous nerve). In order for patients not to know in which group of the study they are included, the probe will be placed on all the aforementioned nerves and they will receive radiofrequency in all of them.

Data will be obtained through the application of questionnaires, for the evaluation of the participants, regarding pain intensity, knee function, analgesic consumption, quality of life and occurrence of adverse effects. The questionnaires will be applied before the block test, to evaluate baseline measurement; after the block test, to verify if there was at least 50% improvement; on the day of the CRF, immediately before the procedure, after the CRF procedure: after 1 week, 1 month, 2 months, 3 months, 4 months, 5 months, and 6 months. For the conservative group, the questionnaires will be applied following the same times established for the intervention groups. The results will be obtained through appropriate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 40 years or older;
* Patients diagnosed with knee OA through X-rays and MRI (Alhback classification 2 or 3);
* Patients with chronic knee pain for more than 3 months at the time of inclusion;
* Patients with moderate to severe knee pain (score of 5 or more on the visual analog scale)
* Patients who are literate, can read and write, and have a good understanding of written and verbal language.

Exclusion Criteria:

* Patients younger than 40 years old, even if diagnosed with knee OA;
* Patients not diagnosed through imaging tests with OA;
* Patients who have undergone previous knee surgery in the last 3 months before inclusion;
* Patients who have received intra-articular corticosteroid injection in the last 3 months before inclusion;
* Patients with uncontrolled neurological or psychiatric disease;
* Patients with uncontrolled diabetes;
* Pregnant patients;
* Cancer diagnosed patients;
* Patients with lumbar radiculopathy;
* Patients on continuous anticoagulant therapy;
* Patients who are not literate, can not read and write, and have not a good understanding of written and verbal language.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Analyze the efficacy of cooled radiofrequency in patients with chronic knee osteoarthritis pain. | 7 months
  Patients will be evaluated regarding pain intensity (by means of the visual analog scale - VAS), knee function (by means of the WOMAC score translated and validated for the Portuguese language), analgesic consumption (by means of the quantitative analgesic questionnaire - QAQ), the patient's quality of life (using the SF-12 questionnaire translated and validated for the Portuguese language), and the occurrence of adverse effects (using the patients' reports) before the block test, to assess the baseline measurement, and after the block test, to check if there was at least a 50% improvement; on the day of the CRF, immediately before the procedure, after the CRF procedure after 1 week, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months.

SECONDARY OUTCOMES:
Analyze the lesions of the neurotomized nerves | 2 months
  After the CRF procedure, patients will undergo MRI. The images will be evaluated for the characterization of the nerve lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela F Rodrigues, Ph.D, Principal Investigator — Universidade Federal de Alfenas; Carlos Marcelo de Barros, MD, FIPP, Study Chair — Sinpain Ltda; Universidade Federal de Alfenas; Ranielly A Andrade, MD, Study Chair — Santa Casa de Alfenas; Lúcio César H Silva, MD,FIPP,CIPS, Study Chair — SINPAIN LTDA; Charles A de Oliveira, MD,FIPP, Study Chair — SINPAIN LTDA; Paulo Renato B da Fonseca, MD,FIPP,MBA, Study Chair — SINPAIN LTDA; Fabrício D Assis, MD,FIPP, Study Chair — SINPAIN LTDA; Tiago S Freitas, MD,Ph.D,FIPP, Study Chair — SINPAIN LTDA; Vanessa BB Marques, Ph.D, Study Director — Universidade Federal de Alfenas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlone AG, Grothaus O, Jacobs C, Duncan ST. Is Cooled Radiofrequency Genicular Nerve Block and Ablation a Viable Option for the Treatment of Knee Osteoarthritis? Arthroplast Today. 2021 Feb 8;7:220-224. doi: 10.1016/j.artd.2020.12.003. eCollection 2021 Feb. PMID 33604437
- [Background] Fonkoue L, Behets CW, Steyaert A, Kouassi JK, Detrembleur C, De Waroux BLP, Cornu O. Accuracy of fluoroscopic-guided genicular nerve blockade: a need for revisiting anatomical landmarks. Reg Anesth Pain Med. 2019 Aug 26:rapm-2019-100451. doi: 10.1136/rapm-2019-100451. Online ahead of print. PMID 31451628
- [Background] Fonkoue L, Behets C, Kouassi JK, Coyette M, Detrembleur C, Thienpont E, Cornu O. Distribution of sensory nerves supplying the knee joint capsule and implications for genicular blockade and radiofrequency ablation: an anatomical study. Surg Radiol Anat. 2019 Dec;41(12):1461-1471. doi: 10.1007/s00276-019-02291-y. Epub 2019 Jul 23. PMID 31338537
- [Background] Fonkoue L, Behets CW, Steyaert A, Kouassi JK, Detrembleur C, De Waroux BL, Cornu O. Current versus revised anatomical targets for genicular nerve blockade and radiofrequency ablation: evidence from a cadaveric model. Reg Anesth Pain Med. 2020 Aug;45(8):603-609. doi: 10.1136/rapm-2020-101370. Epub 2020 Jun 18. PMID 32561652
- [Background] Gonzalez FM. Cooled Radiofrequency Genicular Neurotomy. Tech Vasc Interv Radiol. 2020 Dec;23(4):100706. doi: 10.1016/j.tvir.2020.100706. Epub 2020 Oct 5. PMID 33308582